CLINICAL TRIAL: NCT01907074
Title: Quantitative Liver Function Tests Using Cholates
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 011-063
Record Dates: First submitted 2013-07-22; First posted 2013-07-24 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: End Stage Liver Disease
Keywords: liver function tests; end stage liver disease; cirrhosis; living liver donor
MeSH Terms: conditions — End Stage Liver Disease; Fibrosis | interventions — Cholates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cholates Compound (Experimental)
  Interventions: Drug: Cholates

INTERVENTIONS:
Drug: Cholates — Cholates is given intravenously (IV push) and by mouth, once per study visit

SUMMARY:
As the treatments for liver disease and the availability of liver transplantation have progressed, the number of patients with end stage liver disease continues to increase. This has increased the need to risk-stratify patients with cirrhosis to better direct their treatments and provide an accurate prognosis for their outcomes. The traditional assessment of the liver patient has been limited to imaging, static measures of "liver function tests" and liver biopsy. This protocol is designed to increase the spectrum of tests in the evaluation of the patient with end stage liver disease.

DETAILED DESCRIPTION:
This study involves using the dual cholate test as our quantitative liver function test of choice. Clearance of the oral cholate provides an assessment of portal blood flow. Clearance of the intravenous (IV) cholate provides an assessment of the systemic blood flow. The ratio of these clearances indicates the fraction of cholate that is shunted to the systemic circulation, and is called the cholate shunt fraction.2

This study will measure cholate elimination rate constant (cholate Kelim), clearance of orally administered cholate, clearance of intravenously administered cholate and cholate shunt. This study will compare the presence and extent of the cholate clearances and shunt fraction with the presence and extent of hepatic fibrosis and portal hypertension (as measured by a hepatic venous pressure gradient [HVPG] procedure.)

The patients who will be enrolled in this study may or may not be those who are undergoing clinically indicated hepatic venous pressure gradient (HVPG) measurements at Baylor University Medical Center, with or without a liver biopsy. Patients having the HVPG measurements will be admitted to Baylor University Medical Center (BUMC) and prepared in the routine clinical fashion for their clinically-indicated HVPG measurement. The cholate test, including blood draws, will be performed after the HVPG procedure. The cholate test may also be performed in the Hepatology clinic

ELIGIBILITY:
Inclusion Criteria:

* End-stage liver disease patient or Living Liver Donor or Congenital Heart Disease patients
* Age: 18 yr to 80 yr
* Patients or Legal Authorized Representative (LAR) must provide written consent and be willing and able to adhere to study requirements
* Stage 3-4 fibrosis by METAVIR score or clinical evidence of advanced fibrosis (End-stage liver disease patients only)

Exclusion Criteria:

* Hepatic encephalopathy Grade 3 or 4
* Pregnancy or intent to become pregnant
* Subjects with inability to provide consent for one's self
* Subjects with a life expectancy < 1 year
* Subjects who have participated in an investigational drug study within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-06-23 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness and accuracy of quantitative liver function testing using oral and IV cholate in patients with end-stage liver disease OR in patients who donate a portion of their liver | 1 year

SECONDARY OUTCOMES:
Compare presence and extent of the cholate clearances | One year

OTHER OUTCOMES:
Annual tests to measure changes in liver function | one year

CONTACTS AND LOCATIONS:
Overall Officials: James Trotter, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No